CLINICAL TRIAL: NCT05297396
Title: A Pilot Study of Slow Opioid Tapering Compared to Continued Opioid Therapy in Treating Chronic Non-Cancer Pain
Brief Title: Slow Opioid Tapering Pilot Study of Patients Using Chronic Opioid Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Terrence J. Witt, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-009836
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Opioid Use
Keywords: Chronic opioid therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Slow Tapering of Chronic Opioid Therapy (Experimental): Subjects who are on a stable dose of daily opioid therapy for at least 6 months will have their opioid medication doses slowly and gradually reduced every 4 weeks.
  Interventions: Other: Slow Tapering of Chronic Opioid Therapy
- Continued Opioid Therapy (No Intervention): Subjects who are on a stable dose of daily opioid therapy for at least 6 months will stay on the same dose of opioids they are currently using at the beginning of the study for the entire 12-month duration of the study.

INTERVENTIONS:
Other: Slow Tapering of Chronic Opioid Therapy — Clinically prescribed daily opioids reduced by no more than 10 morphine milligram equivalent per day (MMED) each month for 12 months
  Arms: Slow Tapering of Chronic Opioid Therapy

SUMMARY:
The purpose of this study is to find out if patients who have been taking a stable dose of opioids for chronic pain would experience any worsening pain, quality of life and functioning, as well as symptoms of depression and anxiety if their opioid medications are gradually and very slowly reduced.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide consent.
* Ability to participate in all aspects of this study.
* Using tablet or capsule form of one or two of the designated opioid preparations daily (at least 95% of days) during the previous 6 months, anticipated long term use and no active plans for tapering. Specific opioid preparations designated for inclusion will be based on the frequency of use by patients on the Chronic Opioid Registry as well as tablet or capsule characteristics which allow encapsulation by the Research Pharmacy. Participants who have been prescribed the following oral opioids will be recruited into the study: tramadol 50mg tablet or capsule; hydrocodone-acetaminophen (APAP) 5mg-325mg tablet or capsule; hydrocodone-APAP 7.5mg-325mg tablet or capsule; hydrocodone-APAP 10mg-325mg tablet or capsule; oxycodone 5mg tablet or capsule; oxycodone 10mg tablet or capsule; oxycodone-APAP 5mg-325mg tablet or capsule; oxycodone 10mg-325mg tablet or capsule; morphine sulfate extended release 15mg tablet or capsule; morphine sulfate extended release 30mg tablet or capsule; morphine sulfate immediate release 15mg tablet or capsule; morphine sulfate immediate release 30mg tablet or capsule.
* Primary care provider prescribing chronic opioid therapy within MCHS NW WI and in agreement with patient participation.
* Average daily morphine milligram equivalent (MME) dose at enrollment equal to or less than 90.

Exclusion Criteria:

* Daily or intermittent use of transdermal, liquid, intravenous or intramuscular forms of opioid during the last 6 months.
* Use of methadone or buprenorphine.
* Use of an opioid containing preparation with three or more active ingredients.
* Active cancer treatment, other than non-melanoma dermatological cancers. This includes patients either currently receiving or planning to receive any type of cancer treatment other than hormonal therapy.
* Active or planned pregnancy.
* COT being prescribed for indications other than chronic non-cancer pain (i.e., restless leg syndrome).
* Enrollment in hospice care.
* Active suicidal planning or intent as reported on PHQ9.
* Acquisition of controlled medications from clinicians other than PCP or associated clinicians in the previous 6 months as noted in the Prescription Drug Monitoring Program.
* Use of opioids and/or benzodiazepines other than those prescribed by PCP or associated clinicians, or the use of illicit substances other than THC, as found in urine drug testing within the previous 6 months.
* Known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in measures of quality of life | Baseline, 3 months, 6 months, 9 months, 12 months
  Measured by the Medical Outcomes Study Questionnaire Short Form Health 36 Survey (SF36v2).The SF-36 is a multi-purpose self-reported survey designed to capture adult patients' perceptions of their own health and well-being.

SECONDARY OUTCOMES:
Change in measures of depression | Baseline, 3 months, 6 months, 9 months, 12 months
  Measured using the Physical Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-assessment survey which is a reliable and valid measure of depression severity used in both the clinical and research field. Total scores on a scale of 1-27 with higher score indicated higher depression severity.
Change in measures of anxiety | Baseline, 3 months, 6 months, 9 months, 12 months
  Measured using the Generalized Anxiety Disorder Questionnaire-7 (GAD-7). The GAD-7 is a valid and efficient tool for screening for generalized anxiety disorder and assessing its severity in clinical practice and research. Patients indicate one of the 4 numbers (representing severity) associated with 7 problems. Total score symptom range 0-21 with higher score indicated higher anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Witt, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials